CLINICAL TRIAL: NCT01274884
Title: Prospective Series of Acute Acromioclavicular Dislocations Grade III+. Arthroscopic Fixation With Tightrope (R).
Brief Title: Tightrope Fixation of Acromioclavicular Joint Dislocation - a Prospective Series
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Asker og Baerum (Other)
Responsible Party: Principal Investigator, Wender Figved, MD, PhD, Orthopaedic Surgeon, Sykehuset Asker og Baerum
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACLUX2010
Record Dates: First submitted 2011-01-11; First posted 2011-01-12 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Acromioclavicular Joint Dislocation
Keywords: Acromioclavicular; Injury; Dislocation; Surgery
MeSH Terms: conditions — Wounds and Injuries; Joint Dislocations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acromioclavicular joint dislocation (Active Comparator): Surgery: Arthroscopic repair using the Tightrope fixation device
  Interventions: Procedure: Tightrope fixation

INTERVENTIONS:
Procedure: Tightrope fixation — Arthroscopic repair
  Other Names: Tightrope (R) (Arthrex, Naples, Florida)

SUMMARY:
Several surgical techniques are used for the treatment of acute acromioclavicular joint dislocations. The investigators investigate a new method using arthroscopic repair using the Tightrope fixation device.

DETAILED DESCRIPTION:
The Tightrope consists of a suspension system with a strong suture thread intertwined between an oval button and a round button, which is inserted through drilling holes in the clavicula and the coracoid. The investigators want to prospectively evaluate the results in a series of 25 patients.

ELIGIBILITY:
Inclusion Criteria:

* Acute acromioclavicular joint dislocation
* 18 years or older

Exclusion Criteria:

* Unable to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Constant score | 1 Year
  Shoulder outcome score

SECONDARY OUTCOMES:
Plain radiographs | 1 Year
VAS Pain | 1 Year
  Visual analogue acale 1-10
VAS Satisfaction | 1 Year
  Visual analogue acale 1-10

CONTACTS AND LOCATIONS:
Overall Officials: Wender Figved, MD, PhD, Study Director — Baerum Hospital, Vestre Viken, Norway; Odd A Lien, MD, Principal Investigator — Baerum Hospital, Vestre Viken, Norway
Locations (1):
- Asker and Baerum Hospital, Baerum, Rud, Norway